CLINICAL TRIAL: NCT03465800
Title: Understanding Mechanisms of Exercise Behavior Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-0008
Record Dates: First submitted 2018-02-28; First posted 2018-03-14 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Overweight and Obesity; Physical Activity; Incentives
Keywords: overweight; obesity; physical activity; exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Monitoring (Active Comparator): Participants self-monitor their physical activity
  Interventions: Behavioral: self-monitoring
- Daily Incentives (Experimental): daily payments for physical activity
  Interventions: Behavioral: self-monitoring; Behavioral: daily incentives
- Delayed Lump Sum Incentives (Experimental): lump sum payments for physical activity
  Interventions: Behavioral: self-monitoring; Behavioral: delayed lump sum incentives

INTERVENTIONS:
Behavioral: self-monitoring — self-monitoring of physical activity
Behavioral: daily incentives — daily incentive payments for physical activity
  Arms: Daily Incentives
Behavioral: delayed lump sum incentives — delayed lump sum payments for physical activity
  Arms: Delayed Lump Sum Incentives

SUMMARY:
This research seeks to examine psychological factors that may impact relationship between incentives and health behavior engagement, specifically physical activity. Additionally, it will compare the impact of two different incentive schedules on behavior engagement, one providing immediate rewards (i.e. rewards received on a daily basis) and another providing delayed rewards (i.e. rewards received at the end of the study period), with an active self-monitoring intervention condition in which no rewards are offered. Study participants will provide reports of their physical activity each day for three weeks, and in the two incentive conditions, they will receive small monetary rewards for their physical activity. Following the three week reporting and reward period, participants will complete two additional assessments, measuring psychological constructs and behavior engagement following the cessation of rewards. The study will also examine how cognitive and anthropomorphic factors may contribute to intervention response and the effects on psychological constructs.

ELIGIBILITY:
Inclusion Criteria:

* Complete less than 150 minutes of moderate-vigorous physical activity weekly
* Daily access to the internet for 3 weeks following baseline research visit
* Have or are willing to create an account on PayPal
* Willing to wear a heart rate monitor watch during physical activity for 3 weeks
* BMI greater than or equal to 25, from self-reported height and weight

Exclusion Criteria:

* Diagnosis of cardiovascular, metabolic, or renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Moderate-vigorous physical activity minutes | Week 3
  summed minutes of weekly moderate intensity physical activity & vigorous intensity physical activity
Self-Efficacy for physical activity | Week 3
  8-item self-report scale measuring self-efficacy (Social Cognitive Theory, Bandura, 1977; also called "perceived behavioral control", Theory of Planned Behavior, Ajzen, 1985); scores are a mean of 8 items, scored 1-7 with higher scores indicative of greater self-efficacy
Moderate-vigorous physical activity minutes | Week 5
  summed minutes of weekly moderate intensity physical activity & vigorous intensity physical activity
Self-Efficacy for physical activity | Week 5
  8-item self-report scale measuring self-efficacy (Social Cognitive Theory, Bandura, 1977; also called "perceived behavioral control", Theory of Planned Behavior, Ajzen, 1985); scores are a mean of 8 items, scored 1-7 with higher scores indicative of greater self-efficacy
Attitudes toward physical activity | Week 3
  12-item self-report scale (Theory of Planned Behavior, Ajzen, 1985); scores are a mean of 12 items scored from -5 to +5, with higher scores indicative of more positive attitudes
Attitudes toward physical activity | Week 5
  12-item self-report scale (Theory of Planned Behavior, Ajzen, 1985); scores are a mean of 12 items scored from -5 to +5, with higher scores indicative of more positive attitudes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No